CLINICAL TRIAL: NCT04101786
Title: Kinematic and Electromyographic Analysis of Different Hip Adductors Exercises
Brief Title: Analysis of Different Hip Adductors Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Dean of Faculty, University of Primorska
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP-FVZ-HipAdductorsExercises
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Injury of Hip and Thigh
Keywords: sport; injury; prevention; rehabilitation; groin pain; adductor strain
MeSH Terms: conditions — Hip Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hip adductors exercise variations — The participants will perform different exercise variations targeting hip adductors in randomized order.

SUMMARY:
Groin injuries present a major problem in sports due to its high frequency, long-lasting symptoms and high risk of re-injury. The most common groin injury is the adductor strain (around two thirds of all groin injuries), while the biggest risk factors are previous injury and lower hip adductors strength. The purpose of this study is to present and biomechanically evaluate several new strengthening exercises targeting hip adductors. Exercises will be performed with the use of our novelty device, which enables eccentric strengthening of the hip adductors in different hip and knee positions. We hypothesize that performing modified hip adductors exercises using the novelty device could enable participants to perform hip adduction throughout larger ROM during eccentric contractions, while changing hip and/or knee angle will differently affect muscle activity and produced joint torques. The latter could be helpful for preventive or rehabilitative training for hip adductors strain injuries, in which therapists want to target specific hip adductor muscle.

DETAILED DESCRIPTION:
Following the general warm-up (light aerobic activity, dynamic stretching exercises and bodyweight strength exercises), the electromyographic (EMG) sensors and kinematic markers will be attached to the participant, who will then perform the maximal voluntary contractions for the purpose of EMG normalization. Then the participant will perform new hip adductor exercises using the novelty device, which enables hip adduction eccentric contractions in different hip and knee positions. The latter is important when trying to target specific hip adductor muscle, since different hip and/or knee angles differently affect individual muscle activity and joint torques. Exercises will be performed in randomized order, while the EMG and kinematic signals will be synchronously captured. EMG muscle activity and joint torques, produced during the exercises, will be analysed. Descriptive statistics will be calculated and reported as mean ± standard deviation. Shapiro-Wilk test will be used for testing of normality and Levene's test for equality of variances. Differences among corresponding variables will be obtained from different exercises and tested with the analysis of the variance for repeated measurements. For pair-wise comparisons, paired 2-tailed post-hoc t-tests with Bonferroni's correction will be used. The level of statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Performing regular physical activity, experience with strength training.

Exclusion Criteria:

Neural, muscular, skeletal or connective tissue injuries during the last 12 months in the area of the back, hips and legs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Muscle activity | 3 hours
  Muscle activity of (bilateral) adductor longus, gluteus maximus, gluteus medius, rectus abdominis and obliquus externus will be measured using electromyographic sensors.
Net joint torque | 3 hours
  Net joint torques at the knee and hip will be calculated from kinematic data, measured in frontal plane using 3D kinematic motion capture system.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Principal Investigator — Faculty of health sciences, University of Primorska
Locations (1):
- Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No